CLINICAL TRIAL: NCT06524453
Title: Study on the Safety and Effectiveness of a Rehabilitation Exercise Program for Individuals With Spinal Cord Injury in Community: A Randomized Controlled Trials
Brief Title: Exercise Program for Individuals With SCI in Community
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCI exercise RCT
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries; Exercise Program; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): A 20-session structured rehabilitation exercise program for individuals with SCI
  Interventions: Behavioral: Wheelchair accessible exercise program
- Control group (No Intervention): Maintain their daily lives without any intervention

INTERVENTIONS:
Behavioral: Wheelchair accessible exercise program — 1. Stretching exercise
     * Dynamic and static
     * Neck, shoulder, elbow, wrist, trunk
     * 10 minutes
  2. Aerobic exercise
     * High intensity interval training
     * Arm ergometer or wheelchair running
     * 20 mins
  3. Strengthening exercise
     * Shoulder and chest, elbow joint major muscle; shoulder and trunk stabilization exercise
     * 3 sets of 10
     * 20 minutes
  4. Stretching exercise
     * Dynamic and static
     * Neck, shoulder, elbow, wrist, trunk
     * 10 minutes
  Arms: Exercise group

SUMMARY:
Patients with spinal cord injury (SCI) who have reduced mobility have difficulty exercising on their own without proper guidance in the community. Community-based exercise programs are effective in removing various barriers such as lack of exercise programs, lack of experts, and lack of facilities. This study aims to verify the effectiveness and safety of a systematically designed customized exercise program for patients who live in the community and want to participate in exercise. Our study results will serve as a basis for creating an environment where more individuals with SCI can continue to exercise proactively and in the long term.

DETAILED DESCRIPTION:
People with SCI must perform regular exercise to improve function, quality of life, and reduce medical costs. However, SCI people with reduced mobility have difficulty exercising on their own without proper guidance in the community. Rehabilitation exercise for SCI people should be applied based on accurate functional assessment, and risk factors related to exercise should also be assessed. Community-based exercise programs are effective in removing various barriers such as lack of exercise programs, lack of experts, and lack of facilities.

This study aims to verify the effectiveness and safety of a systematically designed customized exercise program for SCI people who live in the community and want to participate in exercise. Based on the results of many previous studies, the investigators expect that program participants will have improved cardiopulmonary endurance and quality of life. Our study results will serve as a basis for creating an environment where more people with SCI can continue to exercise preemptively and in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients who are 19-65 years old or above and residing in the local community
* Individuals who can not walk independently for more than 10 meters without assistance from others
* Individuals whose elbow extensor strength is greater than muscle manual test (MMT) Fair

Exclusion Criteria:

* Individuals who have difficulty understanding the exercise program or expressing their symptoms
* Individuals who cannot participate in the intervention exercise program due to serious cardiovascular diseases
* Individuals who are deemed unsuitable for this study by a specialist in rehabilitation medicine due to other medical conditions

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
6 minute push test | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Sub-maximal exercise test used to assess aerobic capacity and endurance. Longer distances indicate better athletic ability.

SECONDARY OUTCOMES:
Spinal cord independence measure III | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Tool to evaluate independence of spinal cord injury patients. The total score ranges from 0 to 100, and the higher the score, the more independent the patient is.
Modified functional reach test | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Assessing balance in sitting posture. Measures the maximum distance a person can extend forward while sitting in a fixed posture.
Grip strength | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Force applied by the hand to pull on or suspend from objects. It is widely used to assess sarcopenia and as a surrogate indicator of muscle strength. Measured in kg, the higher the value, the stronger the grip is considered.
Arm curl | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Tests upper limb endurance. Measures the number of times a participant can hold a dumbbell (4kg for men, 2kg for women) for 2 minutes and fully bend and straighten their arms. The higher the number, the better the function and strength.
Back scratch test | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Measures how close the hands can be brought together behind the back. If the fingertips touch then the score is zero. If they do not touch, measure the distance between the finger tips (a negative score), if they overlap, measure by how much (a positive score).
Beck anxiety inventory | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Anxiety measuring tool. Each item is scored 0-3 points, with a total score of 0-63 points. A score of 0-7 indicates minimal anxiety, a score of 8-15 indicates mild anxiety, a score of 16-25 indicates moderate anxiety, and a score of 26-63 indicates severe anxiety.
Beck depression inventory | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Depression measuring tool. Each item is scord 0-3 points, with a total score of 0-63 points. A score of 0-13 indicates minimal depression, a score of 14-19 indicates mild depression, a score of 20-28 indicates moderate depression, and a score of 29-63 indicates severe depression.
Fat-free mass from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  A method used to measure the components of the body. It is the total amount (kg) of body components excluding body fat, and the higher it is, the better the body composition is interpreted.
Fat-free mass index from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  A method used to measure components of the body. This is an indicator that standardizes fat-free mass according to body size. The higher it is, the more muscle mass and the better health.
Percent body fat from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  A method used to measure the components of the body. The normal range varies depending on age and gender. The lower the score within the general normal range, the better the health. The higher it is, the higher the risk of obesity related diseases.
skeletal muscle mass from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  A method used to measure the components of the body. Normal range varies depending on age and gender. The higher it is within the general normal range, the better the health. The lower it is, the higher the risk of lack of strength and sarcopenia.
EuroQol 5 Dimension 5 Level | Baseline evaluation and follow-up evaluation immediately after average 8-weeks of exercise program
  Self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Converting the patient's response results using quality weights has a value between 0.000 and 1.000. A higher score means a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hwa Ko, PhD, Study Chair — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No